CLINICAL TRIAL: NCT01181479
Title: Open-label, Randomized, Parallel Group, Study of Efficacy and Safety of a Transdermal Contraceptive Delivery System (TCDS) in Comparison to a Low-dose Oral Contraceptive Containing 0.02 mg EE and 0.1 mg LNG in a 21-day Regimen.
Brief Title: Study to Evaluate the Contraceptive Efficacy/Safety of a Low Dose EE/LNG Transdermal Contraceptive Delivery System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agile Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATI-CL12; 57731 (Other: FDA)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Contraception
Keywords: Contraceptive
MeSH Terms: interventions — Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AG200-15 (cycles 1-13) (Experimental): AG200-15 containing ethinyl estradiol and levonorgestrel. Type of intervention is drug.
  Interventions: Drug: AG200-15 (cycles 1-13)
- Lessina crossover to AG200-15 (Active Comparator): Lessina containing ethinyl estradiol and levonorgestrel for 6 cycles followed by AG200-15 for 6 cycles. Type of intervention is drug.
  Interventions: Drug: Lessina crossover to AG200-15

INTERVENTIONS:
Drug: AG200-15 (cycles 1-13) — AG200-15 containing ethinyl estradiol and levonorgestrel
  Other Names: transdermal patch
  Arms: AG200-15 (cycles 1-13)
Drug: Lessina crossover to AG200-15 — Low dose oral contraceptive containing 20 mcg ethinyl estradiol and 100 mcg Levonorgestrel in 21 day regimen for 6 cycles followed by AG200-15 for 6 cycles.
  Other Names: hormonal oral contraception and transdermal patch
  Arms: Lessina crossover to AG200-15

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of a low dose transdermal contraceptive delivery system containing ethinyl estradiol and levonorgestrel.

DETAILED DESCRIPTION:
Comparative evaluation of AG200-15 versus OC with regard to safety, contraceptive efficacy, cycle control (bleeding pattern), subject compliance and serum concentrations of EE and LNG. To evaluate TCDS wearability (including adhesion).

ELIGIBILITY:
Inclusion Criteria:

Healthy females

* 17(in states where the legal age of consent to receive contraceptives is 17)-40 years
* Regular, consistent menstrual cycles between 25 and 35 days
* Sexually active women requesting birth control
* In good general health, confirmed by medical history, physical (including gynecologic) examination and screening laboratory values

Exclusion Criteria:

* Known or suspected pregnancy;
* Lactating women
* Significant skin reaction to transdermal preparations or sensitivity to surgical / medical tape
* Any disease that may worsen under hormonal treatment (cardiovascular, liver, metabolic)
* Use of other contraceptive methods than study medication

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1504 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Garner, MD, MPH, Study Director — Agile Therapeutics
Locations (80):
- United States (80):
  - Agile Investigational Site, Huntsville, Alabama
  - Agile Investigational Site, Mobile, Alabama
  - Agile Investigational Site, Chandler, Arizona
  - Agile Investigational Site, Green Valley, Arizona
  - Agile Investigational Site, Tucson, Arizona
  - Agile Investigational Site, Little Rock, Arkansas
  - Agile Investigational Site, La Mesa, California
  - Agile Investigational Site, Los Angeles, California
  - Agile Investigational, Sacramento, California
  - Agile Investigational Site, San Diego, California
  - Agile Investigational Site, Santa Ana, California
  - Agile Investigational Site, Vista, California
  - Agile Investigational Site, West Hills, California
  - Agile Investigational Site, Boulder, Colorado
  - Agile Investigational Site, Colorado Springs, Colorado
  - Agile Investigational Site, Denver, Colorado
  - Agile Investigational Site, Fort Collins, Colorado
  - Agile Investigational Site, Wheat Ridge, Colorado
  - Agile Investigational Site, Milford, Connecticut
  - Agile Investigational Site, New London, Connecticut
  - Agile Investigational Site, Waterbury, Connecticut
  - Agile Investigational Site, Boynton Beach, Florida
  - Agile Investigational Site, Clearwater, Florida
  - Agile Investigational Site, Daytona Beach, Florida
  - Agile Investigational Site, DeLand, Florida
  - Agile Investigational Site, Fort Myers, Florida
  - Agile Investigational Site, Jacksonville, Florida
  - Agile Investigational Site, Pinellas Park, Florida
  - Agile Investigational Site, South Miami, Florida
  - Agile Investigational Site, St. Petersburg, Florida
  - Agile Investigational Site, West Palm Beach, Florida
  - Agile Investigational Site, Atlanta, Georgia
  - Agile Investigational Site, Decatur, Georgia
  - Agile Investigational Site, Sandy Springs, Georgia
  - Agile Investigational Site, Champaign, Illinois
  - Agile Investigational Site, Chicago, Illinois
  - Agile Investigational Site, Indianapolis, Indiana
  - Agile Investigational Site, Newburgh, Indiana
  - Agile Investigational Site, Overland Park, Kansas
  - Agile Investigational Site, Wichita, Kansas
  - Agile Investigational Site, Lexington, Kentucky
  - Agile Investigational Site, Louisville, Kentucky
  - Agile Investigational Site, Marrero, Louisiana
  - Agile Investigational Site, Lincoln, Nebraska
  - Agile Investigational Site, Las Vegas, Nevada
  - Agile Investigational Site, Edison, New Jersey
  - Agile Investigational Site, Lawrenceville, New Jersey
  - Agile Investigational Site, Rochester, New York
  - Agile Investigational Site, Cary, North Carolina
  - Agile Investigational Site, Charlotte, North Carolina
  - Agile Investigational Site, Kernersville, North Carolina
  - Agile Investigational Site, Raleigh, North Carolina
  - Agile Investigational Site, Salisbury, North Carolina
  - Agile Investigational Site, Wilmington, North Carolina
  - Agile Investigational Site, Winston-Salem, North Carolina
  - Agile Investigational Site, Akron, Ohio
  - Agile Investigational Site, Cincinnati, Ohio
  - Agile Investigational Site, Cleveland, Ohio
  - Agile Investigational Site, Columbus, Ohio
  - Agile Investigational Site, Englewood, Ohio
  - Agile Investigational Site, Mayfield Heights, Ohio
  - Agile Investigational Site, Oklahoma City, Oklahoma
  - Agile Investigational Site, Tulsa, Oklahoma
  - Agile Investigational Site, Medford, Oregon
  - Agile Investigational Site, Jackson, Tennessee
  - Agile Investigational Site, Knoxville, Tennessee
  - Agile Investigational Site, Memphis, Tennessee
  - Agile Investigational Site, Austin, Texas
  - Agile Investigational Site, Bedford, Texas
  - Agile Investigational Site, Corpus Christi, Texas
  - Agile Investigational Site, Dallas, Texas
  - Agile Investigational Site, Houston, Texas
  - Agile Investigational Site, San Antonio, Texas
  - Agile Investigational Site, Sugar Land, Texas
  - Agile Investigational Site, Webster, Texas
  - Agile Investigational Site, Salt Lake City, Utah
  - Agile Investigational Site, Newport News, Virginia
  - Agile Investigational Site, Norfolk, Virginia
  - Agile Investigational Site, Richmond, Virginia
  - Agile Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Kaunitz AM, Portman D, Westhoff CL, Mishell DR Jr, Archer DF, Foegh M. New contraceptive patch wearability assessed by investigators and participants in a randomized phase 3 study. Contraception. 2015 Mar;91(3):211-6. doi: 10.1016/j.contraception.2014.11.013. Epub 2014 Nov 25. PMID 25586864
- [Derived] Kaunitz AM, Portman D, Westhoff CL, Archer DF, Mishell DR Jr, Foegh M. Self-reported and verified compliance in a phase 3 clinical trial of a novel low-dose contraceptive patch and pill. Contraception. 2015 Mar;91(3):204-10. doi: 10.1016/j.contraception.2014.11.011. Epub 2014 Nov 25. PMID 25582984
- [Derived] Kaunitz AM, Portman D, Westhoff CL, Archer DF, Mishell DR Jr, Rubin A, Foegh M. Low-dose levonorgestrel and ethinyl estradiol patch and pill: a randomized controlled trial. Obstet Gynecol. 2014 Feb;123(2 Pt 1):295-303. doi: 10.1097/AOG.0000000000000095. PMID 24402597

RESULTS

PARTICIPANT FLOW:
Groups:
- AG200-15 (Cycles 1-13): Intervention with drug: AG200-15 containing ethinyl estradiol and levonorgestrel. Administered for cycles 1-13.
- Lessina (Cycles 1-6): The Lessina regimen was taken for Cycles 1-6.
- Lessina (Cycles 1-6) Crossover to AG200-15 (Cycles 7-13): Intervention with drug: Lessina containing 20 mcg ethinyl estradiol and 100 mcg levonorgestrel in 21 day regimen cycles 1-6 followed by AG200-15 for cycles 7-13.
Period: Subjects Receive AG200-15 or Lessina
Arm/Group | AG200-15 (Cycles 1-13) | Lessina (Cycles 1-6) | Lessina (Cycles 1-6) Crossover to AG200-15 (Cycles 7-13)
Started (Includes all subjects that were randomized.) | 1129 | 375 | 0 (This column is a subset of the Lessina completers in the "Lessina (Cycles 1-6)" column.)
Completed | 485 | 249 | 0
Not Completed | 644 | 126 | 0
Period: Crossover Subjects Recieve AG200-15
Arm/Group | AG200-15 (Cycles 1-13) | Lessina (Cycles 1-6) | Lessina (Cycles 1-6) Crossover to AG200-15 (Cycles 7-13)
Started | 0 | 0 | 249 (This column is a subset of the Lessina completers in the "Lessina (Cycles 1-6)" column.)
Completed | 0 | 0 | 150
Not Completed | 0 | 0 | 99

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- AG200-15: Intervention is drug: AG200-15 containing ethinyl estradiol and levonorgestrel for cycles 1-13.
- Lessina Crossover to AG200-15: Intervention with drug: Lessina containing 20 mcg ethinyl estradiol and 100 mcg levonorgestrel in 21 day regimen cycles 1-6 followed by AG200-15 for cycles 7-13.
- Total: Total of all reporting groups
Arm/Group | AG200-15 | Lessina Crossover to AG200-15 | Total
Number analyzed (Participants) | 1043 | 230 | 1273
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 2 | 7
  Between 18 and 65 years | 1038 | 228 | 1266
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.38 (5.663) | 26.86 (5.738) | 26.46 (5.677)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1043 | 230 | 1273
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1043 | 230 | 1273

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy
Description: Pregnancy outcomes was determine by measuring Pearl index. Pearl Index is the number of on-therapy pregnancies times 1300 divided by the number of 28-day on-therapy cycles and is an estimate of the number of pregnancies per 100 woman-years of product use.
Time Frame: AG200-15: 6 months; Lessina: 6 months; AG200-15: 1 year
Population: Subjects in the Safety population, age 17-35 with a BMI <32, were analyzed.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Groups:
- AG200-15 for Cycle 7-13: Subjects that applied AG200-15 for cycles 7-13.
- Lessina: Subjects that only received Lessina for cycles 1-6.
- AG200-15 for Cycle 1-13: Subjects that applied AG200-15 for all cycles (1-13)
Arm/Group | AG200-15 for Cycle 7-13 | Lessina | AG200-15 for Cycle 1-13
Number analyzed (Participants) | 675 | 220 | 827
Pearl Index | 5.41 [2.35 to 8.46] | 6.67 [0.84 to 12.5] | 6.43 [4.13 to 8.72]

2. Other Pre Specified Outcome: Cycle Control
Description: Measuring the breakthrough bleeding (BTB) and/or breakthrough spotting (BTS). Measured as a percent of total number of cycles in each Arm/Group with BTB and/or BTS.
Time Frame: 6 months
Population: Number of subjects with documented cycle information.
Measure: Number; unit: percentage of cycles with BTB/BTS
Groups:
- AG200-15 for Cycle 1-6: Subjects that applied AG200-15 for cycles 1-6.
Arm/Group | AG200-15 for Cycle 1-6 | Lessina
Number analyzed (Participants) | 715 | 246
percentage of cycles with BTB/BTS | 23.9 | 21.2
Statistical Analysis 1: Comparison: AG200-15 for Cycle 1-6 vs Lessina; Test type: Equivalence — Comparison of AG200-15 and Lessina for cycles 1-6; p = 0.067, Chi-squared

3. Other Pre Specified Outcome: Pharmacokinetics of Levonorgestrel (LNG) and Ethinyl Estradiol (EE)
Description: Measurement of plasma concentrations of LNG and EE for cycles 2, 6 and 13.
Time Frame: Lessina: 6 months; AG200-15: 1 year; AG200-15: 6 months
Population: Subjects that received contraceptive and were analyzed for LNG and EE.
Measure: Mean (95% Confidence Interval); unit: pg/ml
Groups:
- Lessina Cycles 1-6: Subjects that only received Lessina for cycles 1-6.
- AG200-15 for Cycle 1-13: Subjects that applied AG200-15 for cycles 1-13.
- AG200-15 for Cycles 7-13: Subjects switched hormonal contraceptive from Lessina to AG200-15 for cycle 7-13.
Arm/Group | Lessina Cycles 1-6 | AG200-15 for Cycle 1-13 | AG200-15 for Cycles 7-13
Number analyzed (Participants) | 326 | 933 | 144
pg/ml
  EE for cycle 2 | 35.4 [31.9 to 38.8] | 30.5 [29.0 to 32.1] | NA [NA to NA] — Non-applicable because cycle 2 data entered here.
  EE cycle 6 | 40.1 [33.3 to 46.9] | 36.7 [34.3 to 39.0] | NA [NA to NA] — Non-applicable because cycle 6 data entered here.
  EE cycle 13 | NA [NA to NA] — Non-applicable because cycle 13 data entered here. | 31 [28.5 to 33.5] | 33.4 [29.1 to 37.8]
  LNG cycle 2 | 2386 [2180 to 2592] | 1201 [1136 to 1266] | NA [NA to NA] — Non-applicable because cycle 2 data entered here.
  LNG cycle 6 | 2611 [2355 to 2867] | 1753 [1636 to 1871] | NA [NA to NA] — Non-applicable because cycle 6 data entered here.
  LNG cycle 13 | NA [NA to NA] — Non-applicable because cycle 13 data entered here. | 1590 [1452 to 1727] | 1750 [1521 to 1979]

4. Other Pre Specified Outcome: Self-reported Irritation at Application Site
Description: Evaluation of irritation at application site was determined using the following scores:
  0: None
  1. Mild
  2. Moderate
  3. Severe
Time Frame: 1 year
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- All Subjects Who Applied AG200-15: Intervention with drug: AG200-15 containing ethinyl estradiol and levonorgestrel
Arm/Group | All Subjects Who Applied AG200-15
Number analyzed (Participants) | 1273
Score on scale | 1.35 (0.964)

5. Other Pre Specified Outcome: Patch Adhesion by Investigator Evaluation at Each Visit
Description: Evaluation of patch adhesion was determined using the following scores:
  0: >= 90% adhered (no lift)
  1. >= 75% adhered but < 90% (some edges showing lift)
  2. >= 50% adhered but < 75% (half of system lifts off)
  3. < 50% (> half of system lifts off, but undetached)
  4. patch completely detached
Time Frame: 1 year
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Subjects Who Applied AG200-15
Number analyzed (Participants) | 1273
Score on a scale | 0.29 (0.823)

6. Other Pre Specified Outcome: Self-reported Itching at Patch Application Site
Description: Evaluation of itching at patch application site was determined using the following scores:
  0: None
  1. Mild
  2. Moderate
  3. Severe
Time Frame: 1 year
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Subjects Who Applied AG200-15
Number analyzed (Participants) | 1273
Score on a scale | 1.48 (0.948)

ADVERSE EVENTS:
Groups:
- All AG200-15: All subjects that received AG200-15, including subjects that switched from Lessina to AG200-15 for cycles 7-13.
Arm/Group | All AG200-15 | Lessina
All-Cause Mortality (participants affected / at risk) | 0/1273 | 1/344
Serious Adverse Events (participants affected / at risk) | 14/1273 | 4/344
Other Adverse Events (participants affected / at risk) | 484/1273 | 112/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All AG200-15 (N=1273) | Lessina (N=344)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Embolism Venous (Vascular disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastointerstinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All AG200-15 (N=1273) | Lessina (N=344)
Nasopharyngitis (Infections and infestations) | 74 (74) | 12 (12)
Sinusitis (Infections and infestations) | 45 (45) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 51 (51) | 7 (7)
Urinary tract infection (Infections and infestations) | 44 (44) | 11 (11)
Cervical Dysplasia (Reproductive system and breast disorders) | 80 (80) | 17 (17)
Nausea (Gastrointestinal disorders) | 58 (58) | 14 (14)
Human papilloma virus test positive (Investigations) | 40 (40) | 7 (7)
Headache (Nervous system disorders) | 50 (50) | 16 (16)
Vomiting (Gastrointestinal disorders) | 22 (22) | 10 (10)
Dysmenorrhea (Reproductive system and breast disorders) | 20 (20) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Approval by Agile Therapeutics, Inc. of any publication, including oral presentations and abstracts, utilizing data or any information from the ATI-CL12 study is required prior to publication submission.